CLINICAL TRIAL: NCT04371796
Title: Exploratory Efficacy and Safety Study of PD-1 Inhibitor Sintilimab (IBI308) in the Neoadjuvant Treatment of Patients With Resectable II-IIIA NSCLC
Brief Title: Sintilimab (IBI308) in the Neoadjuvant Treatment of Patients With Resectable II-IIIA NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Innovent Biologics, Inc. (Other)
Responsible Party: Principal Investigator, Juan LI, MD, MD, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK2019001
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms; Non-small-cell Lung Cancer
Keywords: NSCLC; neoadjuvant; Sintilimab
MeSH Terms: conditions — Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab injection (Experimental): * Drugs: Eligible patients received two doses of intravenous sintilimab (200 mg) every 3 weeks (Q3W). Each infusion time is 30-60min.
  * Surgery: The patient underwent imaging examinations within 7 days prior to surgery, including chest CT and related metastatic examinations. The patient underwent surgery 6-8 weeks after the first dose.
  Interventions: Drug: Sintilimab injection

INTERVENTIONS:
Drug: Sintilimab injection — Sintilimab injection 200mg, 2cycles of treatment before surgery
  Other Names: IBI308; Xindili Dankang

SUMMARY:
The aim of this study was to investigate the safety and efficacy of Sintilimab (IBI308) in patients with resectable NSCLC, and to provide new treatment options for neoadjuvant therapy in patients with stage II-IIIA NSCLC

DETAILED DESCRIPTION:
Sintilimab injection (IBI308) as neoadjuvant therapy in patients with resectable NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old to 75 years old, male or female;
2. Histologically or cytologically confirmed NSCLC (stage II-IIIA, American Joint Committee on Cancer, eighth edition) that was surgically resectable;
3. Being treatment-naive and the diameter of primary tumor was greater than or equal to 1 cm;
4. ECOG performance status score: 0-1;
5. The function of important organs meets the following requirements (no blood components and cell growth factors are allowed for 2 weeks before the start of study): Absolute neutrophil count (ANC)≥1.5×10 E+9/L; platelets≥100×10E+9/L / L; hemoglobin ≥9g/dL; serum albumin(ALB)≥2.8g/dL; a total bilirubin (TBil) of≤1.5 ULN, ALT and AST≤2.5 ULN, in case of liver metastasis, ALT and AST≤5 ULN; creatinine clearance rate≥ 50mL/min(Cockcroft-Gault);thyroid function is normal.
6. Estimated survival time≥3 months;
7. PD-L1 expression level ≥ 1%；
8. Patients were voluntarily enrolled in the study and signed an informed consent form (ICF) with good adherence and follow-up.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease;
2. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose>10 mg / day of prednisone or other therapeutic hormones);
3. History of interstitial lung disease;
4. Severe allergic reactions to other monoclonal antibodies;
5. Previous allogeneic organ transplantation or hemopoietic stem cell transplantation;
6. Have clinical symptoms or disease that are not well controlled ;
7. Grade III to grade IV congestive heart failure;
8. Uncontrolled hypertension;
9. Artery thrombosis, embolism, or ischemia within 6 months before study treatment;
10. Coagulation disorders;
11. Active and uncontrolled infection;
12. The patient has previously received other PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1;
13. Any other known malignant tumor;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate(MPR)(<10% viable tumor cells) | At time of surgery
  To assess the major pathologic response rate (<10% viable tumor cells) in patients receiving Sintilimab Injection

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 2 years
  the proportion of patients with a best overall response of CR, PR or SD in the whole body, as assessed per RECIST 1.1 by the investigator.
Overall response rate (ORR) | up to 2 years
  the proportion of patients with a best overall confirmed response of CR or PR in the whole body as assessed per RECIST 1.1 by the investigator
Disease-free survival (DFS) | up to 2 years
  Defined as the time from date of surgery until recurrence of tumor or death from any cause
Incidence of irAEs | up to 2 years
  Immune-related AE per Common Terminology Criteria for Adverse Events (CTCAE V5.0)
Incidence of SAEs | up to 2 years
  Grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute

IPD SHARING:
Plan to Share IPD: No